CLINICAL TRIAL: NCT02809339
Title: Improving Quality of Care for Patients With Recurrent Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Other Study IDs: MOGYN24
Record Dates: First submitted 2016-03-07; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-04

CONDITIONS: Ovarian Neoplasms; Quality of Life
Keywords: Chemotherapy; ovarian cancer; Patient reported outcome; Quality of Care
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epithelial ovarian cancer
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires

SUMMARY:
Ovarian cancer is a major cause of cancer related death among women. The disease is usually advanced at diagnosis, because specialist referral is delayed due to vague nature of presenting symptoms. Primary treatment is successful, but most patients experience recurrence. Complaints due to disease and therapy overlap. Furthermore treatment schedules are similar in response rate and survival rates. Toxicity of therapy as scored by the physician is best documented, but varies depending on type of chemotherapy. Moreover most knowledge is acquired in clinical trials and not in daily practice. Patient reported outcome (PROs) concerning effects on symptoms, velocity of relief and quality of life (QoL) by the different regimens is sparce. Also it is unknown which symptoms are best relieved. Most trials take into account progression or survival as primary endpoint but not often symptom relief, which is especially important for patients with recurrent disease, without no chance of cure anymore. Knowledge on rating of problems and needs of patients with recurrent ovarian cancer (ROC) to support them in the course of their disease is needed to come to an evidence based and patient centered treatment of choice together with the patient. Physicians most frequently use the Common Toxicity Criteria (CTC) scale for grading of side effects of treatment, but discrepancies with patient experiences is high. Routine collection of PROs may therefore improve patient expectations and management. In this project the investigators intend to augment knowledge by PROs of different chemotherapy schedules for recurrent ovarian cancer in order to improve shared decision making with the physician.

Objective: primary objective of this project is to explore the relief of symptoms due to ROC, the speed with which this occurs by different chemotherapy schedules and development of complaints due to the regimen of chemotherapy. Secondary the investigators intend (1) to assess preferential symptom relief by patients, (2) to correlate toxicity and symptoms of disease to tumor assessed response to chemotherapy and (3) to correlate symptom relief by psychosocial context.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent EOC or tubal carcinoma or peritoneal carcinoma;
* Histologically and/or cytologically proven epithelial ovarian cancer (including carcinosarcoma of the ovaries)
* Measurable or evaluable disease confirmed by radiological imaging OR ca 125
* ECOG ≤2
* Estimated life expectancy ≥12 weeks
* Patients must be accessible for treatment and follow-up
* Fit to receive chemotherapy

Exclusion Criteria:

* Patients with benign ovarian cancer;
* Patients with non-epithelial cancer;
* Bowel obstruction, sub-occlusive disease or presence of symptomatic brain metastases;
* Patients with other malignancy occurring within 5 years before enrollment
* Patients with impaired cognitive functioning or analphabetic patients
* Patients with an inability to fill in surveys digitally

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with recurrent epithelial ovarian cancer (EOC), tubal carcinoma or peritoneal carcinoma with measurable disease by radiology or tumor-marker and in adequate physical condition (ECOG≤2) to receive chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Velocity of disease symptom relief and its duration by systemic therapy measured by change in MOST questionnaires on PROs and response to therapy | Change in MOST questionnaires as measured before start of therapy, at week 3, 6, 9 and 18 and and there after every 3 months until progression or 1 year

SECONDARY OUTCOMES:
Change in patient reported disease symptoms top 3 due to systemic therapy on their top 3 of complaints | change measured by questionnaire before start of therapy, at week 9 and 18 and at time of progression or 1 year
Change in top 3 complaints due to chemotherapy | change measured by questionnaire before start of therapy, at week 9 and 18 and at time of progression or 1 year
Change in patient reported psychosocial wellbeing | Change measured by HADS questionnaires before start of therapy, at week 9 and 18 and at time of progression or 1 year
Change in patient reported empowerment | Change measured by NEV questionnaire before start of therapy, at week 9 and 18 and at time of progression or 1 year
Change in patient reported needs | Change measured on CASUN questionnaire before start of therapy, at week 9 and 18 and at time of progression or 1 year
Response to therapy by CA-125 (according to GCIG criteria and radiology by RECIST 1.1 criteria) | change measured before start of therapy, at week 9 and 18 and at time of progression or 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nelleke Ottevanger, M.D. PhD, Principal Investigator — Internist - Oncologist and Principal investigator

IPD SHARING:
Plan to Share IPD: Undecided